CLINICAL TRIAL: NCT01515111
Title: Knowledge and Recommendations on Tobacco Cessation and Other Preventive Interventions Among Internal Medicine Staff in Guatemala Teaching Hospitals
Brief Title: Guatemala Internal Medicine Physicians' Knowledge of Non-communicable Disease Clinical Preventive Services
Status: Completed | Type: Observational
Sponsor: Unidad de Cirugía Cardiovascular (Other)
Collaborators: International Development Research Centre, Canada (Other Government); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Juan Enrique Corral, Research Fellow, Unidad de Cirugía Cardiovascular
Other Study IDs: IDRC-006; RITC of IDRC (Other Grant/Funding Number: 105068-002)
Record Dates: First submitted 2012-01-13; First posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Non-communicable Diseases
Keywords: Non-communicable diseases; Preventive services; Medical education; Guatemala
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Internal Medicine Staff: All interns, residents and attendings training (or working) at an Internal Medicine department of a Guatemalan teaching hospital.

SUMMARY:
A national cross-sectional survey was conducted to evaluate recommendations on clinical preventive services and additional information on non-communicable disease prevention. Trained surveyors interviewed interns, residents and attendings of the Internal Medicine departments of all teaching hospitals in Guatemala. Analysis compared recommendation practices within and between hospitals.

DETAILED DESCRIPTION:
A voluntary, anonymous, self-completed, cross-sectional survey was administered to all available internal medicine staff in Guatemalan teaching hospitals.

The questionnaire included: physician's demographics, work time dedicated to outpatients, knowledge of leading causes of death in Guatemala, guidelines used for non-communicable disease prevention, simulated cases asking for recommendation(s) on different preventive services for asymptomatic adults (i.e. whether they recommended them or not, appropriate frequency and starting age, preferred screening method, and availability of the service(s) at their hospital). The survey also assessed barriers faced in providing adequate services, and opinions on who should implement changes in national health care and in medical education.

The answers given by the internal medicine staff were compared with the United States Preventive Services Task Forces (USPSTF) Recommendations and Guatemalan Ministry of Health Guidelines.

Analysis compared recommendation practices within and between hospitals.

ELIGIBILITY:
Inclusion Criteria:

* All interns, internal medicine residents and attendings (including department director, unit directors and regular attendings) that are currently training or working in an Internal Medicine department in any of the ten teaching hospitals in Guatemala.

Exclusion Criteria:

* Staff that is on vacations, on sick leave or suspended by any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Internal medicine interns, residents or attendings of any of the teaching hospitals in Guatemala.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Recommendations of clinical preventive services for non-communicable diseases. | After accepting to participate in the study, participants will be followed the time necesary to complete the structured questionnaire, an average of 1 hour.
  Recommendations on eleven clinical preventive services for non-communicable diseases were evaluated considering:
  * Whether they recommended them or not
  * Appropriate frequency and starting age
  * Preferred screening method
  * Availability of the service(s) at their hospital

SECONDARY OUTCOMES:
Barriers faced in providing adequate services. | After accepting to participate in the study, participants will be followed the time necesary to complete the structured questionnaire, an average of 1 hour.
  Self-perceived barriers to provide clinical preventive services adequately.
Opinion on who should implement changes in clinical preventive services provision. | After accepting to participate in the study, participants will be followed the time necesary to complete the structured questionnaire, an average of 1 hour.
  Participant's opinion on who should be responsible to implement changes in:
  * Chronic disease prevention in national health care
  * Medical education in this field.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Barnoya, M.D. MPH., Study Chair — Unidad de Cirugía Cardiovascular
Locations (10):
- Guatemala (10):
  - Hospital Nacional de Escuintla, Escuintla, Departamento de Escuintla
  - Hospital Universitario Esperanza, Guatemala City, Departamento de Guatemala
  - Hospital Hermano Pedro, Guatemala City, Departamento de Guatemala
  - Hospital Roosevelt, Guatemala City, Departamento de Guatemala
  - Unidad de Cirugía Cardiovascular, Guatemala City, Departamento de Guatemala
  - Hospital Centro Médico Militar, Guatemala City, Departamento de Guatemala
  - Hospital General San Juan de Dios, Guatemala City, Departamento de Guatemala
  - Hospital General de Enfermedad Común - IGSS, Guatemala City, Departamento de Guatemala
  - Hospital Regional de Occidente, San Juan de Dios, Quetzaltenango, Departamento de Quetzaltenango
  - Hospital Nacional Pedro Bethancourt, Antigua Guatemala, Departamento de Sacatepéquez

REFERENCES:
- [Derived] Corral JE, Arnold LD, Argueta EE, Ganju A, Barnoya J. Clinical preventive services in Guatemala: a cross-sectional survey of internal medicine physicians. PLoS One. 2012;7(10):e48640. doi: 10.1371/journal.pone.0048640. Epub 2012 Oct 31. PMID 23119077